CLINICAL TRIAL: NCT07140562
Title: Prospective, Multi-Center, Single-Arm Study: Safety and Technical Feasibility of the Tangent Tricuspid Annular Therapy System for Transcatheter Valve Repair in Patients With Severe, Symptomatic Functional Tricuspid Regurgitation
Brief Title: Safety and Feasibility Study: Transcatheter Valve Repair in Severe Symptomatic Functional Tricuspid Regurgitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tangent Cardiovascular Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-001
Record Dates: First submitted 2025-08-06; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Tricuspid Regurgitation Functional; Tricuspid Regurgitation (TR); Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tangent Tricuspid Annular Therapy System Treatment Group (Experimental): Subjects will receive the experimental device according to the protocol. Primary safety and technical efficacy will be assessed, as well as secondary performance measures.
  Interventions: Device: Tricuspid Annular Therapy System

INTERVENTIONS:
Device: Tricuspid Annular Therapy System — A transcatheter device designed for tricuspid valve repair.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and technical success of the Tangent Tricuspid Annular Therapy System in patients with severe, symptomatic functional tricuspid regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-90 years old at the time of consent
2. Symptomatic functional tricuspid regurgitation (without co-existing degenerative disease) despite being adequately treated with optimal medical therapy by the Local Heart Team for at least 30 days prior to the study consent
3. Severe, massive or torrential functional tricuspid regurgitation, as determined by qualifying transesophageal echocardiogram (TEE) and/or transthoracic echocardiogram (TTE) using the 5-grade classification
4. TEE imaging confirms adequate visualization of valve for TR quantification and procedural guidance
5. The Local Heart Team determines the candidate is suitable for transcatheter tricuspid valve repair
6. Subject or legally authorized representative has provided informed consent and agrees to return for all required post-procedure follow-up visits

Exclusion Criteria:

1. Estimated life expectancy of less than 12 months
2. Systolic pulmonary artery pressure (sPAP) >70 mmHg as assessed by TTE or right heart catheterization
3. Acutely decompensated, defined as hypotension with SBP <90 mmHg, use of hemodynamic support devices or inotropes or uncontrolled arterial hypertension with SBP >180 mmHg within 30 days of the study procedure
4. Severe COPD dependent on home oxygen or chronic home oxygen use
5. Echocardiographic evidence of severe right ventricular dysfunction
6. Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation requiring treatment (prior transcatheter or surgical treatment allowable)
7. Any condition that would interfere with the procedure, such as prior tricuspid valve repair, tricuspid valve leaflet anatomy which may preclude device implantation, pacemaker or Implantable Cardioverter Defibrillator (ICD) leads that would prevent appropriate placement or visualization of implant, Ebstein Anomaly (normal annulus position, but valve leaflets attached to walls and septum of the right ventricle)
8. Tricuspid valve stenosis defined as a tricuspid valve orifice of ≤1.0 cm2 and/or mean gradient of ≥5 mmHg
9. New or untreated right heart chamber and/or superior vena cava intracardiac mass, thrombus, or vegetation
10. Degenerative tricuspid or rheumatic tricuspid valve disease
11. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days of the study procedure
12. Implant or revision of any rhythm management device (CRT or CRT-D, ICD, or leadless pacemaker) within 90 days prior to the study procedure
13. Known need for emergent, urgent, or planned surgery or intervention within 30 days following the study procedure, or planned or scheduled cardiac surgery within 12 months following the study procedure
14. Stroke or other major cerebrovascular event within 90 days prior to the study procedure
15. Untreated clinically significant coronary artery disease requiring revascularization, recent (within 30 days of the study procedure) acute coronary syndrome or myocardial infarction
16. Active or recent GI bleed within 30 days prior to the study procedure, or patients contraindicated for oral anticoagulation therapy
17. Bleeding disorders including thrombocytopenia (platelet count <70,000 mm3) or thrombocytosis (platelet count >700,000 mm3)
18. Transfusion-dependent chronic anemia with Hb <9/dL
19. Current or planned pregnancy within 12 months of the study procedure for women of childbearing potential
20. Active or recent endocarditis within 90 days of the study procedure, or sepsis/other systemic infection requiring oral or intravenous antibiotics within 30 days of the study procedure
21. Prior tricuspid repair or tricuspid replacement or prosthetic implant that would interfere with successful deployment or functioning of the Tangent Implant
22. Participation in another pre-market investigational device study or investigational drug study (for a cardiac-related drug)
23. Presence of other anatomic or co-morbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's availability to participate in the clinical investigation or to comply with follow-up requirements
24. Any patient considered to be vulnerable
25. Left ventricular ejection fraction (LVEF) <30%
26. Deep vein thrombosis or pulmonary embolism within 6 months of the study procedure
27. Child-Pugh C cirrhosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Proportion of Patients Free From Device or Procedure-Related Major Adverse Events (MAEs) Through 30-Days Post-Procedure | 30 days post-procedure
  Freedom from device or procedure-related major adverse events (MAEs) through 30 days post-procedure, including:
  * Cardiovascular mortality
  * Stroke
  * Myocardial infarction
  * Major cardiac structural complications
  * Device-related pulmonary embolism (PE)
  * Severe bleeding defined by MVARC
  * Unplanned tricuspid valve re-intervention (percutaneous or surgical)
Primary Technical and Efficacy Endpoint - Measure 1: Technical Success at Completion of the Procedure | At completion of the index procedure
  Technical success upon completion of the procedure in the catheterization lab or operating room, defined as:
  1. Successful delivery and removal of the Delivery System;
  2. Device implanted in the patient as intended.
Primary Technical and Efficacy Endpoint - Measure 2: Procedural Technical Success and TR ≤Moderate at Hospital Discharge | At hospital discharge following the index procedure
  Procedural success at discharge, defined as:
  1. Achieved technical success;
  2. TR classification of moderate or less

SECONDARY OUTCOMES:
Secondary Endpoint - NYHA Functional Class at 30, 90, 180, and 365-Days Post-Procedure | 30 days (±7 days); 90 days (±30 days); 180 days (±30 days); 365 days (±60 days)
  Change from baseline at 30-, 90-, 180-, and 365-days post-procedure in the following:
  a) New York Heart Association (NYHA) functional class
Secondary Endpoint - KCCQ at 30, 90, 180, and 365-Days Post-Procedure | 30 days (±7 days); 90 days (±30 days); 180 days (±30 days); 365 days (±60 days)
  Change from baseline at 30-, 90-, 180-, and 365-days post-procedure in the following:
  b) KCCQ
Secondary Endpoint - 6MWT at 30, 90, 180, and 365-Days Post-Procedure | 30 days (±7 days); 90 days (±30 days); 180 days (±30 days); 365 days (±60 days)
  Change from baseline at 30-, 90-, 180-, and 365-days post-procedure in the following:
  c) 6-minute walk test
Secondary Endpoint - Tricuspid Regurgitation at 30, 90, 180, and 365-Days Post-Procedure | 30 days (±7 days); 90 days (±30 days); 180 days (±30 days); 365 days (±60 days)
  Change from baseline at 30-, 90-, 180-, and 365-days post-procedure in the following:
  d) Tricuspid regurgitation

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay